CLINICAL TRIAL: NCT05540067
Title: Improving Mental Health Among the LGBTQ+ Community Impacted by the COVID-19 Pandemic
Brief Title: Improving Mental Health Among the LGBTQ+ Community
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022003397; RF1MH132348 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Anxiety; Depression
Keywords: Anxiety; Depression; LGBTQ+; COVID-19; Brief intervention; Social support; Acceptance-based behavior therapy
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a 2-arm RCT.
Who Masked: Outcomes Assessor
Masking Description: Blinded raters will conduct interviewer-rated assessments of anxiety and depression (primary outcomes)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acceptance-Based Behavior Therapy (ABBT) (Experimental): The 2-session ABBT will be delivered remotely or in-person, depending on preference.
  Interventions: Behavioral: Acceptance-Based Behavior Therapy (ABBT)
- Treatment-as-Usual (TAU) (Other): Control participants will receive the currently recommended best practices of care at the recruitment site.
  Interventions: Other: Treatment-as-Usual (TAU)

INTERVENTIONS:
Behavioral: Acceptance-Based Behavior Therapy (ABBT) — In the first session, the interventionist will introduce the concept of acceptance and its possible benefits in the context of life values and participant-identified challenges related to the COVID-19 pandemic, mental health, and social support. Interventionists will help participants identify potential challenges to acceptance. At the second session, participants will practice acceptance-based coping skills and a social support behavioral plan will be developed. These discussions will help the participant clarify how best to align their values with decisions on how to manage their mental health and social support in the context of the COVID-19 pandemic.
  Arms: Acceptance-Based Behavior Therapy (ABBT)
Other: Treatment-as-Usual (TAU) — TAU includes brief mental health screening, consultation with providers, and referrals to psychotherapy and/or psychiatric medication.
  Arms: Treatment-as-Usual (TAU)

SUMMARY:
The overall aim of this program of research is to improve the mental health of people who identify as LGBTQ+ by increasing their social support through a brief intervention. The purpose of the proposed project is to establish the effectiveness of our empirically-supported, brief acceptance-based behavioral therapy (ABBT). To achieve the specific aims, the investigators will conduct a fully-powered, randomized clinical trial (n=240) with two treatment arms: treatment-as-usual (TAU) vs. ABBT.

DETAILED DESCRIPTION:
During the COVID-19 pandemic, up to 81% of adults in the United States experienced worsening mental health. A major cause was the social isolation triggered by the pandemic due to quarantining, loss of family or friends, and loss of work. For individuals who lost social connections or were unable to adapt to maintain their connections, social support decreased and loneliness worsened, putting them at much higher risk for anxiety and depressive symptoms.

Importantly, people who identify as LGBTQ+ have been particularly affected by the social isolation caused by the pandemic and were already at much higher risk of social isolation, loneliness, and mental illness, including suicidality, before the pandemic. The objective of this R01 fully-powered trial is to examine the effectiveness of a brief acceptance-based behavioral telehealth intervention (ABBT) to improve mental health during the COVID-19 pandemic by strengthening social support among LGBTQ+ individuals.

The aims of this proposal are: (1) to examine the effectiveness of ABBT in reducing mental health morbidity by conducting a fully-powered, RCT (n=240) of ABBT vs. Treatment-as-Usual; and, (2) to examine potential mediators and moderators of ABBT treatment effects. Primary outcomes will be anxiety and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Present to recruitment clinic for any type of clinical care
* Identify as LGBTQ+
* Self-reported ≥ mild anxiety and/or depressive symptoms, based on the GAD-7 and PHQ-9
* 18 years or older
* Ability to speak and read English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | 39 weeks
  The interviewer-rated HAM-A is a measure of anxiety symptom severity.
Quick Inventory of Depressive Symptomatology - Clinician Rating (QIDS-C) | 39 weeks
  The interviewer-rated QIDS-C is a measure of depressive symptom severity.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | 39 weeks
  The GAD-7 is a self-report measure of anxiety severity.
Patient Health Questionnaire-9 (PHQ-9) | 39 weeks
  The PHQ-9 is a self-report measure of depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Moitra, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share data via The National Institute of Mental Health Data Archive (NDA).
Time Frame: Data will be uploaded to NDA semi-annually. Consistent with NIMH guidelines, there will be no specific time limit regarding how long IPD are available.
Access Criteria: Request to access the data will be evaluated by the MPIs to ensure that they meet reasonable standards of scientific integrity.
URL: http://nda.nih.gov/

REFERENCES:
- [Derived] Moitra E, Brick LA, Cancilliere MK, Elwy AR, Erbe AM, Fenn N, Nunn AS, Salhaney P, Chan PA. A randomized trial of acceptance-based behavioral therapy to improve mental health outcomes for LGBTQ+ persons: Study protocol. Contemp Clin Trials. 2023 Jul;130:107211. doi: 10.1016/j.cct.2023.107211. Epub 2023 May 3. PMID 37146874